CLINICAL TRIAL: NCT01517360
Title: Pharmacological Approach to Improve the Outcome of Social Cognition Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: National Alliance for Research in Schizophrenia and Affective Disorders (Unknown)
Responsible Party: Principal Investigator, Stephen R Marder, MD, Director, VA Desert Pacific Mental Illness Research, Education, and Clinical Center, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Promise # 0041
Record Dates: First submitted 2012-01-19; First posted 2012-01-25 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Social Cognition; Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo+Social Cognitive Skills Training (Active Comparator): The training utilizes skill building techniques that are commonly used in psychiatric rehabilitation. These include breaking down complex social cognitive processes into their components and automating these skills through repetition and practice. The training programs will include 12 sessions and will be administered in a small group format (6-8 participants per group) twice a week for 6 weeks. The treatment groups will include individuals who are assigned to placebo. Each training session will last for about 90 minutes (1 hour training and 30 minutes between placebo administration and start of training).
  Interventions: Other: Placebo; Behavioral: Social Cognitive Skills Training
- Oxytocin+Social Cognitive Skill Training (Experimental): The training utilizes skill building techniques that are commonly used in psychiatric rehabilitation. These include breaking down complex social cognitive processes into their components and automating these skills through repetition and practice. The training programs will include 12 sessions and will be administered in a small group format (6-8 participants per group) twice a week for 6 weeks. The treatment groups will include individuals who are assigned to oxytocin. Each training session will last 90 minutes (1 hour training and 30 minutes between oxytocin administration and start of training).
  Interventions: Drug: Oxytocin; Behavioral: Social Cognitive Skills Training

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 40 IU, intranasal inhalation
  Other Names: Syntocinon
  Arms: Oxytocin+Social Cognitive Skill Training
Other: Placebo — Placebo, matched to Oxytocin, intranasal inhalation
  Arms: Placebo+Social Cognitive Skills Training
Behavioral: Social Cognitive Skills Training — The training utilizes skill building techniques that are commonly used in psychiatric rehabilitation. These include breaking down complex social cognitive processes into their components and automating these skills through repetition and practice. The training programs will include 12 sessions and will be administered in a small group format (6-8 participants per group) twice a week for 6 weeks. Each training session will last for about 90 minutes (1 hour training and 30 minutes between drug administration and start of training).

SUMMARY:
This study will evaluate whether oxytocin will facilitate the learning of social cognitive skills in schizophrenia patients who receive 12 sessions of Social Cognitive Skills Training (SCST). The primary hypothesis is that schizophrenia subjects who are treated with oxytocin will demonstrate greater improvements in a summary measure of social cognition than subjects treated with placebo over the course of SCST.

DETAILED DESCRIPTION:
Individuals with schizophrenia often have serious deficits in their abilities to perceive and interpret socially relevant information. These deficits in social cognition can lead to misunderstanding the intentions of others and failing to interpret social signals that are important for successful social interactions. The relationship between social cognition and functioning has led our group to develop a research agenda that includes understanding the neural underpinnings of social cognitive deficits, measuring these impairments using brain-based biomarkers and clinical assessments, and enhancing our Social Cognitive Skills Training program to improve social cognition and promote recovery.

Oxytocin, which is a hormone and neurotransmitter, is believed to impact social cognition through increased orienting toward and attending to socially salient visual features. There is also evidence that oxytocinergic signaling is impaired in schizophrenia. With this research, we hope to learn whether administration of oxytocin will improve different aspects of social cognition by examining the effects of oxytocin versus placebo administered intranasally before each of 12 sessions of a social cognitive skills training program on measures of independent living, work and social functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders 4th edition
* Stable on an antipsychotic medication
* No change in antipsychotic dose of >10% during the past 3 months

Exclusion Criteria:

* Unable to provide informed consent
* History of epilepsy
* Active medical conditions that would make the study unsafe
* History of serious head injury
* History of hyponatremia

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Composite Social Cognition Score | Baseline, 6 weeks, and 10 weeks
  We will assess emotion management, emotion perception, social context processing/social perception, theory of mind, attributional bias, and empathic accuracy. The primary summary measure for each test will be mean-centered and standardized to create a Z-score that will be averaged to create a single composite score for social cognition, serving as the primary outcome measure. Parallel follow-up analyses will be conducted on individual components to determine which measures are most affected by treatment. Similar secondary analyses will be employed for the event related potential (ERP) and basic cognition measures.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marder, MD, Principal Investigator — Department of Veterans Affairs, University of California Los Angeles
Locations (1):
- West Los Angeles VA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Marder SR, Wirshing WC, Mintz J, McKenzie J, Johnston K, Eckman TA, Lebell M, Zimmerman K, Liberman RP. Two-year outcome of social skills training and group psychotherapy for outpatients with schizophrenia. Am J Psychiatry. 1996 Dec;153(12):1585-92. doi: 10.1176/ajp.153.12.1585. PMID 8942455
- [Background] Horan WP, Kern RS, Tripp C, Hellemann G, Wynn JK, Bell M, Marder SR, Green MF. Efficacy and specificity of social cognitive skills training for outpatients with psychotic disorders. J Psychiatr Res. 2011 Aug;45(8):1113-22. doi: 10.1016/j.jpsychires.2011.01.015. Epub 2011 Mar 4. PMID 21377168
- [Background] Heinrichs M, von Dawans B, Domes G. Oxytocin, vasopressin, and human social behavior. Front Neuroendocrinol. 2009 Oct;30(4):548-557. doi: 10.1016/j.yfrne.2009.05.005. Epub 2009 Jun 6. PMID 19505497
- [Background] Feifel D, Macdonald K, Nguyen A, Cobb P, Warlan H, Galangue B, Minassian A, Becker O, Cooper J, Perry W, Lefebvre M, Gonzales J, Hadley A. Adjunctive intranasal oxytocin reduces symptoms in schizophrenia patients. Biol Psychiatry. 2010 Oct 1;68(7):678-80. doi: 10.1016/j.biopsych.2010.04.039. Epub 2010 Jul 7. PMID 20615494